CLINICAL TRIAL: NCT06143345
Title: High-Intensity Interval Training for Individuals With Isolated Impaired Fasting Glucose: A Proof-of-Concept Study
Brief Title: HIIT in Isolated IFG: A Proof-of-Concept Study
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Due to operational issues
Sponsor: Emory University (Other)
Collaborators: National Center for Advancing Translational Sciences (NCATS) (NIH)
Responsible Party: Principal Investigator, Sathish Thirunavukkarasu, Assistant Professor, Emory University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: STUDY00005855; UL1TR002378 (NIH)
Record Dates: First submitted 2023-11-16; First posted 2023-11-22 (Actual); Last update posted 2026-02-09 (Actual); Status verified 2026-02

CONDITIONS: Isolated Impaired Fasting Glucose
Keywords: Prediabetes; Obesity; High-intensity interval training; Isolated impaired fasting glucose
MeSH Terms: conditions — Prediabetic State; Obesity | interventions — High-Intensity Interval Training; Continuous Glucose Monitoring

STUDY DESIGN:
Who Masked: Outcomes Assessor
Masking Description: Staff conducting the outcome assessments will be blinded to the participants' treatment status.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention Group (Experimental): Intervention participants will complete 24 supervised high-intensity interval training (HIIT) sessions over 8 weeks, with 3 sessions per week on alternate days. Each HIIT session will consist of a 5-minute warm-up, followed by an interval-based workout phase that includes steady up-tempo cadences, sprints, and climbs, interspersed with recovery periods. The session will conclude with a 5-minute cooldown. The workout sessions will initially last 20 minutes and will progressively increase in time based on participants' tolerance and instructor recommendations. Intensity will start at 75% of the estimated maximal heart rate reserve and will increase by 5% weekly, as tolerated and/or deemed necessary by the instructor, over the 8-week intervention period. Participants will receive instructions to maintain a eucaloric diet throughout the study.
  Interventions: Behavioral: High-intensity interval training and eucaloric diet; Device: Continuous glucose monitoring (CGM) (Dexcom G6 Pro CGM sensor)
- Control Group (Active Comparator): Control participants will be instructed to refrain from engaging in intense physical activities during the study period. They will also receive instructions to maintain a eucaloric diet throughout the study.
  Interventions: Behavioral: No intense physical activity and eucaloric diet; Device: Continuous glucose monitoring (CGM) (Dexcom G6 Pro CGM sensor)

INTERVENTIONS:
Behavioral: High-intensity interval training and eucaloric diet — Intervention participants will complete 24 supervised high-intensity interval training (HIIT) sessions over 8 weeks, with 3 sessions per week on alternate days. Each HIIT session will consist of a 5-minute warm-up, followed by an interval-based workout phase that includes steady up-tempo cadences, sprints, and climbs, interspersed with recovery periods. The session will conclude with a 5-minute cooldown. The workout sessions will initially last 20 minutes and will progressively increase in time based on participants' tolerance and instructor recommendations. Intensity will start at 75% of estimated maximal heart rate reserve and will increase by 5% weekly, as tolerated and/or deemed necessary by the instructor, over the 8-week intervention period. Participants will receive instructions to maintain a eucaloric diet throughout the study.
  Other Names: HIIT intervention
  Arms: Intervention Group
Behavioral: No intense physical activity and eucaloric diet — Control participants will be instructed to refrain from engaging in intense physical activities during the study period. They will also receive instructions to maintain a eucaloric diet throughout the study.
  Arms: Control Group
Device: Continuous glucose monitoring (CGM) (Dexcom G6 Pro CGM sensor) — The continuous glucose monitoring (CGM) system comprises a sensor, a transmitter, and a receiver. The sensor measures interstitial fluid glucose levels every 5 minutes, and the transmitter wirelessly sends this glucose data to the receiver. Both intervention and control participants will wear the CGM device in a blinded mode for 10 days before starting the intervention, throughout the 8-week intervention period, and for 10 days post-intervention.
  Other Names: Dexcom G6 Pro CGM sensor

SUMMARY:
This pilot randomized controlled trial will involve 34 physically inactive adults aged 35-65 years with overweight or obesity and isolated impaired fasting glucose (i-IFG). The study aims to assess the feasibility of recruiting and retaining participants, implementing study procedures, and evaluating the acceptability of a high-intensity interval training (HIIT) intervention. Additionally, it will investigate the preliminary efficacy of HIIT in reducing fasting plasma glucose levels and addressing the pathophysiology of i-IFG.

DETAILED DESCRIPTION:
This 1:1 proof-of-concept randomized controlled trial (RCT) will involve 34 physically inactive adults aged 35-65 years who are overweight or obese and have isolated impaired fasting glycemia (i-IFG). Potentially eligible individuals identified through Emory's MyChart electronic health care records system will undergo initial screening via phone calls. Individuals meeting the eligibility criteria will be invited to the Georgia Clinical and Translational Science Alliance at Emory University Hospital in Atlanta for further assessment. During their visit, participants will complete questionnaires, undergo an oral glucose tolerance test, and provide blood samples for insulin. Individuals identified with i-IFG will be randomized into the intervention or control groups.

Individuals assigned to the intervention group will participate in supervised high-intensity interval training (HIIT) sessions using stationary Spin cycle ergometers, in groups of five or fewer. They will wear continuous glucose monitoring (CGM) devices for 10 days before the intervention, throughout the 8-week intervention period, and for 10 days post-intervention. The intervention will be conducted three times a week for eight weeks at the Aerobic Exercise Laboratory in the Rehabilitation Hospital at Emory University. Control participants will be instructed to refrain from engaging in intense physical activities during the study period and will also wear CGM devices for the same duration. All participants will receive instructions to maintain a eucaloric diet throughout the study.

At baseline and after eight weeks, all participants will undergo physical measurements (anthropometrics, blood pressure, and body composition) as well as biochemical measurements (glucose and insulin levels). Additionally, participants in the intervention group will be invited to participate in qualitative in-depth interviews both before and after the HIIT intervention and will complete an intervention acceptability questionnaire upon completion.

The primary outcomes include feasibility metrics, measures of intervention feasibility, acceptability, and appropriateness, and participants' experiences, perceptions, and satisfaction with the HIIT intervention, as well as facilitators and barriers to participation. Secondary outcomes include: 1) Between-group differences in changes from baseline to 8 weeks in mean fasting plasma glucose and insulin levels, indices of β-cell function and insulin resistance, and physical measurements; and 2) CGM metrics: a) Between-group differences in the proportion of time and mean time spent in nocturnal (00:00-06:00) [58] normoglycemia (60 to <100 mg/dl) during the 8-week intervention period and the 10 days following the intervention; b) Within-participant differences in the proportion of time and mean time spent in nocturnal (00:00-06:00) normoglycemia (60 to <100 mg/dl) between exercise and non-exercise days during the 8-week intervention period.

ELIGIBILITY:
Inclusion criteria:

1. Males and females aged 35-65 years
2. Any race or ethnicity
3. BMI ≥25 kg/m2 (≥23 kg/m2 if Asian decent)
4. Physically inactive (<150 min of moderate-intensity or <75 min of vigorous-intensity aerobic physical activity/week)
5. Will be residing in the same location until completion of the study
6. Isolated impaired fasting glucose on the OGTT: FPG 100-125 mg/dl and 2-hr plasma glucose <140 mg/dl

Exclusion criteria:

1. History of diabetes
2. Regular exercise training in the past 6 months
3. Enrolled in weight loss programs in the past 6 months
4. Following a specific diet (e.g., ketogenic, Mediterranean)
5. Pregnant women
6. Breastfeeding
7. Smokers
8. Taking medications known to affect glucose tolerance (e.g., steroids)
9. Taking beta-blockers and calcium channel blockers
10. Taking weight loss medications
11. Underwent bariatric surgery
12. Anemia
13. History of chronic illnesses (e.g., stroke)

Individuals satisfying the eligibility criteria will undergo an OGTT (0, 30, 120 min), and those diagnosed with i-IFG (FPG 100 or 110-125 mg/dl and 2-hr PG <140 mg/dl) will be recruited to the study.

Ages: 35 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2026-06-01 (Estimated); Primary Completion 2026-12-30 (Estimated); Study Completion 2026-12-30 (Estimated)

PRIMARY OUTCOMES:
Response rate in % | Baseline
  No. of individuals responded to the invitation/No. of individuals invited.
Screening yield in % | Baseline
  No. of individuals diagnosed with i-IFG/No. of individuals screened.
Enrolment rate in % | Baseline
  No. of individuals enrolled/No. of individuals diagnosed with i-IFG.
Time to enrollment (mins) | Baseline
  Average time taken from sending the invitation to enrolling one participant in the trial.
Intervention compliance in % | 8 weeks
  No. of HIIT sessions attended/Total no. of HIIT sessions.
Program costs (USD) | From baseline to 8 weeks
  Includes screening cost, cost of procedures, intervention cost, participant incentives, and other costs.
Staff time (mins) | From baseline to 8 weeks
  Time spent screening and recruiting participants, time spent delivering the intervention, time spent making phone calls to participants, time spent implementing the study procedures, and time spent on baseline and follow-up assessments.
Retention rate in % | 8 weeks
  No. of participants attended follow-up visits/No. of participants enrolled.
Feasibility of Intervention Measure (FIM) score | 8 weeks
  The FIM scale will evaluate the feasibility of the intervention, encompassing questions regarding its implementability, possibility, doability, and ease of use. Responses to the questions in the questionnaire will be recorded on a Likert scale of 1 to 5. The mean total score will be calculated by combining the individual Likert points. Higher scores on the FIM scale indicate greater intervention feasibility.
Theoretical Framework of Acceptability (TFA) score | 8 weeks
  The acceptability of the intervention will be assessed through the Theoretical Framework of Acceptability (TFA) questionnaire, which explores affective attitude, burden, ethicality, perceived effectiveness, intervention coherence, self-efficacy, opportunity costs, and general acceptability.
Intervention Appropriate Measure (IAM) score | 8 weeks
  The Intervention Appropriate Measure (IAM) will evaluate the appropriateness of the intervention, including questions about its fittingness, suitability, applicability, and alignment with participants' needs.

SECONDARY OUTCOMES:
Fasting plasma glucose (mg/dl) | 8 weeks
  Change in fasting plasma glucose from baseline to 8 weeks will be compared between study groups.
Fasting insulin (µU/ml) | 8 weeks
  Change in fasting insulin from baseline to 8 weeks will be compared between study groups.
Weight in kg | 8 weeks
  Weight will be measured using a digital weighing scale (Welch Ally-Scale-Tronix, NY, USA) with precision to the nearest 0.1 kg. The change in weight from baseline to 8 weeks will be compared between the intervention and control groups.
BMI in kg/m2 | 8 weeks
  Change in BMI from baseline to 8 weeks will be compared between study groups.
Waist circumference in cm | 8 weeks
  Change in waist circumference from baseline to 8 weeks will be compared between study groups.
Waist-to-hip ratio | 8 weeks
  Change in waist-to-hip ratio from baseline to 8 weeks will be compared between study groups.
Systolic blood pressure in mmHg | 8 weeks
  Change in systolic BP from baseline to 8 weeks will be compared between study groups.
Diastolic blood pressure in mmHg | 8 weeks
  Change in diastolic BP from baseline to 8 weeks will be compared between study groups.
Insulinogenic index (IGI) | 8 weeks
  IGI is a measure of early-phase insulin secretion.
Oral Disposition Index (DIO) | 8 weeks
  DIO is a measure of ß-cell function.
Homeostatic Model Assessment of ß-cell function (HOMA-B) | 8 weeks
  HOMA-B is a measure of ß-cell function.
Matsuda index | 8 weeks
  Matsuda index is a measure of insulin resistance.
Homeostatic Model Assessment of Insulin Resistance (HOMA-IR) | 8 weeks
  HOMA-IR is a measure of insulin resistance.
Hepatic Insulin Resistance Index (HIRI) | 8 weeks
  HIRI is a measure of hepatic insulin resistance.
Muscle Insulin Sensitivity Index (MISI) | 8 weeks
  MISI is a measure of muscle insulin resistance.
Fat percent (%) | 8 weeks
  Fat percent will be obtained by bioimpedance analysis.
Fat mass (kg) | 8 weeks
  Fat mass will be obtained by bioimpedance analysis.
Muscle mass (kg) | 8 weeks
  Muscle mass will be obtained by bioimpedance analysis.
Visceral adipose tissue mass (kg) | 8 weeks
  Visceral adipose tissue mass will be obtained by bioimpedance analysis.
CGM metric: Proportion of time spent in nocturnal (00:00-06:00) normoglycemia (60 to <100 mg/dl) | From baseline to 8 weeks
  Proportion of time spent in nocturnal (00:00-06:00) normoglycemia (60 to <100 mg/dl) during the 8-week intervention period.
CGM metric: Proportion of time spent in nocturnal (00:00-06:00) normoglycemia (60 to <100 mg/dl) | 10 days following the intervention
  Proportion of time spent in nocturnal (00:00-06:00) normoglycemia (60 to <100 mg/dl) during the 10 days following the intervention.
CGM metric: Mean time spent in nocturnal (00:00-06:00) normoglycemia (60 to <100 mg/dl) | From baseline to 8 weeks
  Mean time spent in nocturnal (00:00-06:00) normoglycemia (60 to <100 mg/dl) during the 8-week intervention period.
CGM metric: Mean time spent in nocturnal (00:00-06:00) normoglycemia (60 to <100 mg/dl) | 10 days following the intervention
  Mean time spent in nocturnal (00:00-06:00) normoglycemia (60 to <100 mg/dl) during the 10 days following the intervention.

CONTACTS AND LOCATIONS:
Overall Officials: Sathish Thirunavukkarasu, PhD, Principal Investigator — Emory University

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Thirunavukkarasu S, Ziegler TR, Weber MB, Staimez L, Lobelo F, Millard-Stafford ML, Schmidt MD, Venkatachalam A, Bajpai R, El Fil F, Prokou M, Kumar S, Tapp RJ, Shaw JE, Pasquel FJ, Nocera JR. High-Intensity Interval Training for Individuals With Isolated Impaired Fasting Glucose: Protocol for a Proof-of-Concept Randomized Controlled Trial. JMIR Res Protoc. 2025 Feb 20;14:e59842. doi: 10.2196/59842. PMID 39977858